CLINICAL TRIAL: NCT00262886
Title: Non-Myeloablative HLA-Matched Sibling Allogeneic Peripheral Blood Stem Cell Transplantation for Metastatic Renal Cell Carcinoma
Brief Title: Donor Peripheral Stem Cell or Bone Marrow Transplant in Treating Patients With Relapsed or Refractory Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000449939; URCC-U1801; URCC-RSRB-09084
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Antilymphocyte Serum; Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: graft-versus-tumor induction therapy
Biological: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: A peripheral stem cell transplant or bone marrow transplant from a brother or sister may be an effective treatment for kidney cancer.

PURPOSE: This phase II trial is studying how well a donor peripheral stem cell or bone marrow transplant works in treating patients with relapsed or refractory metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of nonmyeloablative sibling allogeneic peripheral blood stem cell transplantation in patients with relapsed or refractory metastatic renal cell carcinoma.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a pilot study.

* Conditioning regimen: Patients receive cyclophosphamide IV on days -7 and -6 and fludarabine IV on days -5 to -1. Patients receiving 5/6-mismatched cells also receive anti-thymocyte globulin IV on days -5 to -3.
* Allogeneic peripheral blood stem cell (PBSC) infusion: Patients undergo allogeneic PBSC or bone marrow transplantation on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive oral mycophenolate mofetil twice daily on days 0-30. Patients receive tacrolimus IV continuously or orally twice daily beginning on day -2 and continuing up to day 44-100 in the absence of GVHD.
* Donor lymphocyte infusion: Patients with partial or complete T-cell chimerism receive up to 3 donor lymphocyte infusions in the absence of GVHD or progressive disease.

After completion of study treatment, patients are evaluated periodically for 3 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell carcinoma

  * Relapsed or refractory disease
  * Tumor not amenable to complete surgical resection
* No bone metastases only
* No untreated brain metastases
* Measurable disease
* Available sibling donor who is HLA-identical or who has a mismatch at a single HLA locus (i.e., a 6/6 or 5/6 match at the HLA-A, -B, and -DR loci)

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin < 3 mg/dL

Renal

* Creatinine < 2 mg/dL
* No untreated hypercalcemia

Cardiovascular

* LVEF ≥ 40%

Pulmonary

* DLCO ≥ 40%

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test
* HIV-1 and -2 negative
* No uncontrolled infection
* No other active malignancy except basal skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* At least 15 days since prior treatment for renal cell carcinoma
* No other concurrent anticancer therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2001-08; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Response rate based on tumor measurements at 1 year

SECONDARY OUTCOMES:
Toxicity as measured by NCI CTC at days 0, 7, 14, 21 and 28 after transplantation and monthly for 11 months
Overall and disease-free survival at day 100 and 1 year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: J. J. Ifthikharuddin, MD, Principal Investigator — James P. Wilmot Cancer Center; Jane L. Liesveld, MD, Principal Investigator — James P. Wilmot Cancer Center
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States